CLINICAL TRIAL: NCT02220569
Title: PhysioFlow Use in Longterm Screening and Evaluation of Cardiotoxicity in Chemotherapy
Brief Title: PhysioFlow to Detect Cardiotoxicity in Chemo
Acronym: PULSE-ECCho
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nathaniel Bouganim, Dr. Nathaniel Bouganim, Medical Oncologist at Royal Victoria Hospital muhc, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 4073
Record Dates: First submitted 2014-08-14; First posted 2014-08-20 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Chemotherapy, Cancer, Cardiotoxicity, Physioflow
MeSH Terms: conditions — Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
PULSE-ECCho will focus on trying to detect cardiotoxicity in cancer patients receiving chemotherapy early on in order to avoid irreversible damage. In addition to that, we will test if the PhysioFlow is non-inferior to the conventional MUGA scan.

DETAILED DESCRIPTION:
Our objective is to compare the PhysioFlow to the MUGA scan and see if the results are statistically the same using both techniques. This is what is known as a non-inferior study. The advantage of PhysioFlow is that it is non-invasive, fast and it is done at the bedside or while the patient is receiving his or her chemotherapy.

The patient will be tested with the MUGA scan, as per the standard of care, before chemotherapy is initiated and at every 3 months. The patient will also be tested with the PhysioFlow at the same dates of the MUGA scan. In addition to that, the patients will be tested at each chemotherapy cycle with the PhysioFlow.

Should the PhysioFlow indicate the patient has a cardiac toxicity as the patient is receiving chemotherapy, the results will be confirmed with the MUGA scan.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years old
2. Histologically confirmed diagnosis of cancer
3. ECOG 0 to 2
4. Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained
5. Able to adhere to the study visit schedule and other protocol requirements

Control Group

1. Age above 18 years old
2. No previous history of cancer
3. ECOG 0 to 2
4. Did not receive chemotherapeutic agents (even if outside the context of cancer)
5. Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained
6. Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Age less than 18 years
2. ECOG 3-4
3. Suspected or proven severe aortic insufficiency
4. Patient under cardiopulmonary bypass assistance (I.e.: Left ventricular assisting device)
5. Congenital cardiac deformities ,such as septal defects
6. Refuse to comply with the specified visit schedules and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the oncology day clinic at Royal Victoria hospital and receiving chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
comparing the change in ejection fraction measured by physioflow and MUGA scan | at initial diagnosis and after 3 month

SECONDARY OUTCOMES:
acceptance score on the five-point Likert Scale to measure tolerability | up to 24 hrs
  At the end of physioflow and or MUGA scan, a questionnaire to assess acceptance was proposed to all patients. The following aspects were evaluated: preparation and information before the imaging examination, degree of preceding concern, comfort, helplessness during the examination, pain experienced, degree of overall satisfaction. Evaluation was performed with a five-point qualitative Likert scale: very low, low, moderate, high, very high

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Bouganim, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - McGill university health center, Royal Victoria hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec